CLINICAL TRIAL: NCT06785974
Title: Statins to Prevent Immune Checkpoint Inhibitor-induced PRogression of AtherosLerosis
Acronym: SPIRAL
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Jorie Versmissen, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 11670
Record Dates: First submitted 2024-12-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Atherosclerosis; Melanoma; Immune-related Adverse Event
Keywords: Statin; Immune Checkpoint Inhibitor
MeSH Terms: conditions — Atherosclerosis; Melanoma | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention/ Atorvastatin arm (Experimental): Patient will receive 20mg of atorvastatin daily together with ICI-therapy
  Interventions: Drug: Atorvastatin
- Placebo arm (Placebo Comparator): Patient will receive placebo daily together with ICI-therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Daily 20mg atorvastatin.
  Other Names: Lipitor; Atorvastatin Mylan
  Arms: Intervention/ Atorvastatin arm
Drug: Placebo — Daily Placebo in combination with ICI-therapy
  Arms: Placebo arm

SUMMARY:
The goal of this interventional study is to test whether atorvastatin prevents accelerated progression of atherosclerosis in melanoma patients who receive immune checkpoint inhibitor (ICI) therapy. The main questions it aims to answer are:

* difference in percentage growth of total atherosclerotic plaque volume (+ calcified and non-calcified plaque volume) in the descending thoracic segment of the aorta
* difference in percentage growth of total atherosclerotic plaque volume (+ calcified and non-calcified plaque volume) in coronary arteries.

Researchers will compare patients that receive ICI-therapy and atorvastatin with patients that receive ICI-therapy + placebo to see if atorvastatin will prevent accelerated ICI induced plaque growth.

DETAILED DESCRIPTION:
Rationale: Immune checkpoint inhibitors (ICIs) are often highly effective anti-cancer therapies but predispose patients receiving this treatment to cardiovascular disease and thrombotic events. One of the mechanisms by which ICIs increase cardiovascular risk is by stimulation of inflammation and atherosclerosis. Statins (e.g., atorvastatin) are frequently prescribed and effective anti-atherogenic agents, which could provide protective effects on the cardiovascular system in this patient population whilst and after receiving ICI, minimizing cardiovascular sequelae.

The objective of this study is to study if addition of atorvastatin prevents accelerated progression of atherosclerosis during ICI therapy. In addition, the investigators would like to study the effects of atorvastatin during ICI therapy on endothelial function, epicardial fat volume, and hemostatic and inflammatory parameters.

The main study endpoint is the difference in percentage growth of total atherosclerotic plaque volume in the descending thoracic segment of the aorta between intervention and control group, expressed in indexed percentage growth /year.

Secondary endpoints are differences in non-calcified and calcified plaque volume in the thoracic arteries and coronary arteries, epicardial fat volume, endothelial function, and quality of life. Exploratory endpoints include effect on hemostatic and inflammation markers, lipid levels, progression free survival, event free survival, and overall survival.

Trial design Placebo controlled prospective randomised controlled trial.

Trial population Melanoma patients who are scheduled to receive ICI therapy (nivolumab, pembrolizumab, or a combination of anti-PD1/ipilimumab; (neo)adjuvant, irresectable or metastasized melanoma) according to standard-of-care who are also eligible to initiate statin therapy.

The intervention group receives atorvastatin 20mg daily together with ICI therapy. The control group receives placebo together with ICI therapy.

Both groups will undergo two coronary and thoracic CT-scans. In addition, blood withdrawal will take place fourthly during the study. Furthermore, endothelial function will be assessed by means of the EndoPAT device at baseline and after one year of follow-up.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks: Patients in the intervention group will receive atorvastatin, of which safety and tolerability will be carefully monitored. Coronary atherosclerosis will be assessed via two coronary CT-scans, yielding a total limited extra radiation exposure of 4-10mSv. Blood withdrawal will be combined with regular blood withdrawal time points for standard care or will be withdrawn from the intravenous catheter for ICI administration. Vascular endothelial dysfunction will be assessed via Endothelial Peripheral Arterial Tonometry (EndoPAT) by recording finger arterial pulsatile volume change. This non-invasive method forms a minimal extra burden for participating patients. The investigators hypothesize that atorvastatin prevents accelerated progression of atherosclerosis and ameliorates ICI-induced vascular endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria:
* Age ≥ 18 years
* Able to understand the written information and able to give informed consent
* Melanoma diagnosis with planned ICI treatment according to standard of care (nivolumab, pembrolizumab, monotherapy or combination therapy with ipilimumab)
* Presence of atherosclerosis in the descending thoracic aorta at baseline.

Exclusion Criteria:

* Pregnancy or lactation
* Baseline statin use or previously reported statin intolerance
* Current or recent (≤1 year) history of alcohol or drug abuse
* Contra-indication for statin therapy, including:

  * Active liver disease, including ALT/AST levels ≥ 3x ULN
  * (History of) myopathy Congenital muscular disorder History of (drug-induced) rhabdomyolysis History of drug-induced myopathy with elevated creatine kinase (CK)
  * Severe kidney failure (creatinine clearance < 30 ml/min)
* Use of essential medication with (potential) interactions with atorvastatin, including:

  * strong CYP3A4 inhibitors such as clarithromycin, ciclosporin, itraconazol, ketoconazole, voriconazol, posconazol, HCV agents, HIV protease inhibitors
  * BCRP inhibitors such as elbasvir and grazoprevir
  * Fibrates (including gemfibrozil)
* Life expectancy < 12 months
* High MESA-score at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Percentual annual growth of atherosclerotic plaques in the descending thoracic aorta | 1 year
  The percentage difference in atherosclerotic plaque volume in the descending part of the thoracic after 1 year of ICI-therapy will be compared to the atherosclerotic plaque volume at baseline.

SECONDARY OUTCOMES:
Difference in percentage increase in non-calcified and calcified atherosclerotic plaque volume in the descending thoracic aorta | 1 year
  Difference in percentage increase in non-calcified and calcified atherosclerotic plaque volume in the descending thoracic aorta 1 year after the start of ICI therapy in the intervention versus the control group
Difference in percentage increase in total, non-calcified and calcified coronary artery atherosclerotic plaque volume | 1 year
  Difference in percentage increase in total, non-calcified and calcified coronary artery atherosclerotic plaque volume
Difference in increase in coronary calcification score (Agatston score) and Multi-Ethnic Study of Atherosclerosis (MESA) score | 1 year
  Difference in increase in coronary calcification score (Agatston score) and MESA score. MESA score calculates the 10-year risk in percentage of developing coronary heart disease.
Difference in change in epicardial fat volume | 1 year
  Difference in change in epicardial fat volume
Difference in reactive hyperaemia in-dex | 1 year
  Difference in reactive hyperaemia in-dex as a marker of endothelial dysfunc-tion using peripheral arterial tonometry (EndoPAT) between intervention and control group.
Difference in Quality of Life between intervention and control group using the FACT-M and EQ5D5L questionnaire. | Baseline, 3 months, 6 months and 1 year after the start of ICI therapy
  Difference in QoL between intervention and control group using the FACT-M and the EQ5D5L questionnaires
Differences in the number of adverse events | 1 year
  Differences in the number of adverse events between intervention and control group during the first year after start of ICI therapy, graded according to CTCAE criteria, version 5.0.

OTHER OUTCOMES:
The effect of atorvastatin on median Progression Free Survival in months | 1 and 3 years
  The median progression free survival (PFS) in patients with advanced melanoma will be obtained after one and three years and will be calculated in months.
  Progression Free Survival (PFS) is defined as duration from randomization until disease progression.
The effect of statins on the median Overall Survival in months | 1 and 3 years
  The effect of statins on the median overall survival in months in patients with advanced disease after 1 and after 3 years. Overall Survival (OS) is defined as the duration from randomization until death from any cause
The effect of statins on the median Event Free Survival in months | 1 and 3 years
  The effect of statins on the median Event Free Survival in months in patients with advanced disease after 1 and after 3 years. Event Free Survival (EFS) is defined as the time from the start of the study treatment to the occurrence of progression to unresectable melanoma before surgery (in the neoadjuvant setting), disease recurrence, or death due to melanoma or due to treatment, whichever occurs first.
Difference in various concentration levels of hemostatic biomarkers | Baseline, 3 months, 6 months and 1 year after the start of ICI therapy
  Difference in change in concentration levels of various markers of the hemostatic system activation (including d-dimer, fibrinogen, factor VIII, von Willebrand factor) between the intervention and control group at 3 months, 6 months, and 1 year after the start of ICIs.
Difference in serum concentration of cardiovascular risk profile biomarkers | Baseline, 3 months, 6 months and 1 year after the start of ICI therapy
  Difference in serum levels of the following parameters: HsCRP, VCAM, ICAM, TNF-α, IL-1β, IL-6, IL-10, Lipid profile, lp(a) between the intervention and control group at 3 months, 6 months and 1 year after the start of ICIs.

CONTACTS AND LOCATIONS:
Overall Officials: Jorie Versmissen, MD,PhD, Principal Investigator — Department Internal Medicine, Hospital Pharmacy, Erasmus MC Rotterdam
Locations (1):
- Erasmus Universitair Medisch Cetrum Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data will only become available after the study has been completed for at least 1 year. Only the IPD that have given informed consent to use the anonymous data will be available.
  After completion of the study, the Erasmus MC policy for requesting data will be applied. Furthermore, the General Data Protection Regulation must be complied with at all times.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 2 years inclusion, 1 year after completion, 1 year analysis approximately 01-08-2028. Data will be available for 15 years after date of obtaining.
Access Criteria: The data will only become available after the study has been completed for at least 1 year.
  After completion of the study, the Erasmus MC policy for requesting data will be applied. Furthermore, the General Data Protection Regulation must be complied with at all times.

REFERENCES:
- See also: Maarten van der Weijden Foundation — https://www.mvdwfoundation.nl/ondersteunde-projecten/verminderen-van-hart-en-vaatziekte-bij-immunotherapie